CLINICAL TRIAL: NCT01235195
Title: Phase 1, Open-Label, Randomized, Single-Dose, 2-Treatment, 2-Period Crossover Bioequivalence Study Comparing Sertraline Hydrochloride 50 mg Film-Coated Tablets To Sertraline Hydrochloride 50 mg Hard Capsules Under Fasted Conditions
Brief Title: A Study Comparing the Drug Exposure in Humans After Administration of a 50 mg Tablet of Sertraline Hydrochloride as Compared to a 50 mg Capsule of Sertraline Hydrochloride Under Fasted (Nonfed) Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0501097
Record Dates: First submitted 2010-11-03; First posted 2010-11-05 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: bioequivalence study; sertraline 50 mg; capsules vs tablets
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertraline 50 mg capsules (Active Comparator)
  Interventions: Drug: sertraline hydrochloride
- Sertraline 50 mg tablet (Active Comparator)
  Interventions: Drug: sertraline hydrochloride

INTERVENTIONS:
Drug: sertraline hydrochloride — 50 mg capsule, single-dose
  Other Names: Zoloft
  Arms: Sertraline 50 mg capsules
Drug: sertraline hydrochloride — 50 mg tablet, single-dose
  Other Names: Zoloft
  Arms: Sertraline 50 mg tablet

SUMMARY:
This study is designed to determine differences in drug exposure in subjects after being administered 50 mg tablets of sertraline hydrochloride as compared to drug exposure after administering 50 mg capsules of sertraline hydrochloride under fasted (nonfed) conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501097&StudyName=A%20study%20comparing%20the%20drug%20exposure%20in%20humans%20after%20administration%20of%20a%2050%20mg%20tablet%20of%20sertraline%20hydrochloride%20as%20compared%20to%20a%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline 50 mg Capsule, Then Sertraline 50 mg Tablet: Sertraline Hydrochloride 50 milligram (mg) hard gelatin capsule in the first intervention period, Sertraline Hydrochloride 50 mg Film-Coated Tablet in the second intervention period
- Sertraline 50 mg Tablet, Then Sertraline 50 mg Capsule: Sertraline Hydrochloride 50 mg film-coated tablet in the first intervention period, Sertraline Hydrochloride 50 mg hard gelatin capsule in the second intervention period
Period: First Intervention
Arm/Group | Sertraline 50 mg Capsule, Then Sertraline 50 mg Tablet | Sertraline 50 mg Tablet, Then Sertraline 50 mg Capsule
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout Period of At Least 8 Days
Arm/Group | Sertraline 50 mg Capsule, Then Sertraline 50 mg Tablet | Sertraline 50 mg Tablet, Then Sertraline 50 mg Capsule
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Sertraline 50 mg Capsule, Then Sertraline 50 mg Tablet | Sertraline 50 mg Tablet, Then Sertraline 50 mg Capsule
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Entire study population receiving Sertraline Hydrochloride 50 mg as either hard gelatin capsule or film-coated tablet
Arm/Group | Entire Study Population
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to 72 Hours [AUC (0-72)]
Description: AUC (0-72)= Area under the plasma concentration versus time curve from time zero (pre-dose) to 72 hours (0-72).
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants: all treated participants with at least one sertraline concentration were evaluated for pharmacokinetics.
Measure: Mean (Standard Deviation); unit: nanogram hour per milliliter (ng*h/mL)
Groups:
- Sertraline 50 mg Hard Gelatin Capsule: All participants receiving Sertraline Hydrochloride 50 mg Hard Gelatin Capsule
- Sertraline 50 mg Film-Coated Tablet: All participants receiving Sertraline Hydrochloride 50 mg Film-Coated Tablet
Arm/Group | Sertraline 50 mg Hard Gelatin Capsule | Sertraline 50 mg Film-Coated Tablet
Number analyzed (Participants) | 30 | 30
nanogram hour per milliliter (ng*h/mL) | 419.9 (147.14) | 442.1 (169.20)
Statistical Analysis 1: Comparison: Sertraline 50 mg Hard Gelatin Capsule vs Sertraline 50 mg Film-Coated Tablet; Natural log-transformed AUC (0-72) analyzed using a mixed effect model with sequence, period, treatment as fixed effects; subject within sequence as a random effect. Estimates of adjusted mean differences (Test minus Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model. Adjusted mean differences and 90% CIs for differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test divided by Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio (%) of adjusted means = 104.86, 90% CI 2-sided [100.12 to 109.83] — Reference treatment=Sertraline hydrochloride 50 mg hard gelatin capsule. Test treatment=sertraline hydrochloride 50 mg film-coated tablet

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sertraline 50 mg Hard Gelatin Capsule | Sertraline 50 mg Film-Coated Tablet
Number analyzed (Participants) | 30 | 30
nanogram per milliliter (ng/mL) | 17.96 (5.0438) | 19.03 (6.3319)
Statistical Analysis 1: Comparison: Sertraline 50 mg Hard Gelatin Capsule vs Sertraline 50 mg Film-Coated Tablet; Natural log-transformed Cmax analyzed using a mixed effect model with sequence, period, treatment as fixed effects; subject within sequence as a random effect. Estimates of adjusted mean differences (Test minus Reference) and corresponding 90% CIs were obtained from the model. Adjusted mean differences and 90% CIs for differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test divided by Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio (%) of adjusted means = 105.34, 90% CI 2-sided [98.46 to 112.69] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants.
Measure: Median (Full Range); unit: hours
Arm/Group | Sertraline 50 mg Hard Gelatin Capsule | Sertraline 50 mg Film-Coated Tablet
Number analyzed (Participants) | 30 | 30
hours | 5.00 [3.00 to 8.00] | 5.00 [2.00 to 8.00]

4. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Sertraline 50 mg Hard Gelatin Capsule | Sertraline 50 mg Film-Coated Tablet
Number analyzed (Participants) | 30 | 30
ng*h/mL | 471.4 (189.86) | 493.8 (204.90)
Statistical Analysis 1: Comparison: Sertraline 50 mg Hard Gelatin Capsule vs Sertraline 50 mg Film-Coated Tablet; Natural log-transformed AUC (0-∞) analyzed using a mixed effect model with sequence, period, treatment as fixed effects; subject within sequence as a random effect. Estimates of adjusted mean differences (Test minus Reference) and corresponding 90% CIs were obtained from the model. Adjusted mean differences and 90% CIs for differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test divided by Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio (%) of adjusted means = 106.1, 90% CI 2-sided [100.16 to 112.39] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Residual Area Under the Concentration Time Curve [AUC(Res%)]
Description: AUC(res%) is the residual AUC defined as (AUCinf minus AUClast) divided by AUCinf. AUCinf is the area under the plasma concentration-time curve from time zero extrapolated to infinite time. AUClast is the area under the plasma concentration-time curve from zero to the last measured concentration.
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Population: This parameter was not analyzed. It is reported individually for each subject and not analyzed statistically.
Arm/Group | Sertraline 50 mg Hard Gelatin Capsule | Sertraline 50 mg Film-Coated Tablet
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sertraline 50 mg Hard Gelatin Capsule | Sertraline 50 mg Film-Coated Tablet
Number analyzed (Participants) | 30 | 30
hours | 25.45 (3.9067) | 25.40 (3.3831)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sertraline 50 mg Hard Gelatin Capsule | Sertraline 50 mg Film-Coated Tablet
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 11/30 | 13/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline 50 mg Hard Gelatin Capsule (N=30) | Sertraline 50 mg Film-Coated Tablet (N=30)
Palpitations (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Eructation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 2
Catheter site haematoma (General disorders) | 1 | 1
Catheter site swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.